CLINICAL TRIAL: NCT04567849
Title: Decreasing ED Utilization by Nudging Patients to Call Their Provider or Triage Nurse After Women's Health Procedures
Brief Title: Decreasing ED Utilization by Nudging Patients to Call Their Providers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Geisinger Clinic (Other)
Responsible Party: Principal Investigator, Amir Goren, Program Director, Behavioral Insights Team, Geisinger Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2020-0849
Record Dates: First submitted 2020-09-23; First posted 2020-09-29 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Emergency Treatment; Telephone Hotlines
Keywords: Behavioral Economics; Patient Portal

STUDY DESIGN:
Intervention Model Description: Throughout the study, patients will be randomized equally across all three arms.
Who Masked: Participant, Care Provider
Masking Description: Participants (i.e., patients) will not be informed specifically of their assignment to different arms throughout the study. Providers will not be randomized to study arms or informed of patient assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): No intervention control group
- Nudge: call provider (Experimental): This group will receive a patient portal message the morning after completing their procedure. The message will encourage patients to call their recent Women's Health provider (with appropriate phone number listed) if any questions or concerns arise about their healthcare.
  Interventions: Behavioral: message; Behavioral: provider
- Nudge: call tele-nurse (Experimental): This group will receive a patient portal message the morning after completing their procedure. The message will encourage patients to call Geisinger's nurse triage hotline (with appropriate phone number listed) if any questions or concerns arise about their healthcare.
  Interventions: Behavioral: message; Behavioral: tele-nurse

INTERVENTIONS:
Behavioral: message — patient portal message
  Arms: Nudge: call provider; Nudge: call tele-nurse
Behavioral: provider — nudging calling the patient's provider
  Arms: Nudge: call provider
Behavioral: tele-nurse — nudging calling the tele-nurse
  Arms: Nudge: call tele-nurse

SUMMARY:
In the present study, patients will be sent a message shortly after completing a medical procedure that informs or reminds them that they can reach out to Geisinger, and how to do it, if they have any medical issues or concerns. Researchers will assess if such messages make patients more likely to contact Geisinger with post-procedure medical concerns and decrease emergency department utilization.

DETAILED DESCRIPTION:
Decreasing emergency department (ED) over-utilization is a priority for healthcare systems across the country. Patients uncertain about a medical issue routinely end up in the ED when less costly and time-consuming alternatives could have addressed their concern. If patients reach out to healthcare facilities rather than heading directly to the ED, they can often be directed toward resources better suited to their concerns than the ED.

Geisinger is thus working to encourage patients to contact healthcare providers if any concerns arise and patients are uncertain about where to go for care. Patients who have recently had a medical procedure may be particularly valuable to encourage, as they routinely have concerns related to the procedure and discharge can serve as a useful touch-point to remind the patient where they can go for questions or concerns.

In the present study, patients will be sent a patient portal message shortly after completing any Women's Health medical procedure. The message will inform or remind patients how they can reach Geisinger if they have any medical issues or concerns. The purpose of this study is to assess if such messages make patients more likely to contact Geisinger with medical concerns and, in turn, decrease unnecessary ED utilization. This study will A/B test 2 messages, encouraging patients to either call their recent provider directly or to call a tele-nurse hotline, and will assess if these messages perform better than a control group that will not be sent any such message.

Generalized linear models will examine the primary study outcomes as a function of the study arms (between-subjects).

ELIGIBILITY:
Inclusion Criteria:

* Patient had a procedure in Women's Health within the study period (including both surgical and in-office procedures as well as baby delivery)
* Patient is enrolled in myGeisinger, Geisinger's patient portal

Exclusion Criteria:

* If procedure was labor that resulted in fetal demise or stillborn.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11546 (Actual)
Dates: Start 2021-11-16 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
Phone calls | 18 months or as long as it takes to reach N=17,300, whichever occurs first
  Proportion of patients who call the tele-nurse or their provider within 30 days of their appointment
ED utilization | 18 months or as long as it takes to reach N=17,300, whichever occurs first
  Proportion of patients who visit the ED within 30 days of their appointment

SECONDARY OUTCOMES:
Phone calls | 12 months
  Proportion of patients who call the tele-nurse or their provider within 30 days of their appointment
ED utilization | 12 months
  Proportion of patients who visit the ED within 30 days of their appointment
Phone calls - surgical patients only | 18 months or as long as it takes to reach N=17,300, whichever occurs first
  Proportion of patients who call the tele-nurse or their provider within 30 days of their appointment
ED utilization - surgical patients only | 18 months or as long as it takes to reach N=17,300, whichever occurs first
  Proportion of patients who visit the ED within 30 days of their appointment
Phone calls - surgical patients only | 12 months
  Proportion of patients who call the tele-nurse or their provider within 30 days of their appointment
ED utilization - surgical patients only | 12 months
  Proportion of patients who visit the ED within 30 days of their appointment

CONTACTS AND LOCATIONS:
Overall Officials: Amir Goren, PhD, Principal Investigator — Geisinger Clinic
Locations (1):
- Geisinger, Danville, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Data with no personally identifiable information will be made available to other researchers on the Open Science Framework for transparency.
Supporting Information: Analytic Code
Time Frame: The data will become available after publication of study results in a scientific journal and will be available as long as the Open Science Framework hosts the data.
Access Criteria: The data on the Open Science Framework will be open to anyone requesting that information.
URL: http://osf.io

DOCUMENTS (1):
  • Statistical Analysis Plan (2022-03-25): https://cdn.clinicaltrials.gov/large-docs/49/NCT04567849/SAP_000.pdf